CLINICAL TRIAL: NCT01308710
Title: Endothelial Assessment of Risk From Lipids in Youth: Mediterranean Diet
Brief Title: The Effects of a Mediterranean Diet in Pediatric Hyperlipidemia
Acronym: EARLYMedit
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Vanderbilt University (Other); Tufts University (Other); University of Guelph (Other); University of L'Aquila (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: R56NR004909
Record Dates: First submitted 2011-03-03; First posted 2011-03-04 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Hyperlipidemia
Keywords: endothelial function; lipids; pediatrics
MeSH Terms: conditions — Hyperlipidemias | interventions — Fatty Acids, Omega-3; Eicosapentaenoic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acid (Eicosapentaenoic acid) — 1.0 grams daily for 6 weeks
  Other Names: PlusEPA

SUMMARY:
Children with high cholesterol levels are especially vulnerable and are at high risk for early onset coronary heart disease (CHD). Endothelial dysfunction, the earliest phase of CHD, is present in children with elevated cholesterol levels as early as 8 years of age. The long term objective of this study is to develop dietary interventions for the prevention and treatment of endothelial dysfunction in children with common lipid disorders including familial hypercholesterolemia (FH) and familial combined hyperlipidemia (FCH). Increasing evidence suggests that the Mediterranean diet and ω-3 fatty acids found in fish have cardioprotective effects. The specific aims of the study are to: determine whether a Mediterranean diet alone or combined with ω-3 fatty acid (eicosapentaenoic acid)improves endothelial function; evaluate the effects of the dietary interventions on lipids and lipoprotein subclasses; evaluate the effects of the dietary interventions on biomarkers for oxidative stress and inflammation. This study is a randomized, double-blind, placebo-controlled clinical trial that includes 34 children (ages 8-17) treated with the Mediterranean diet and ω-3 fatty acid supplements. A dietary educational behavioral intervention will be conducted over 6 months with individual counseling and group sessions. Endothelial function will be measured noninvasively by high resolution ultrasound of the brachial artery at baseline, 6, 12, 18 and 24 weeks. This study is unique because it is a new intervention designed for children at high risk for early CHD with a dietary component and supplementation with ω-3 fatty acids. If effective, this intervention would be broadly applicable in the community and lend valuable insight about dietary therapy to prevent the progression of CHD in hyperlipidemic children.

ELIGIBILITY:
Inclusion Criteria:

* Children (8-17 years old)
* Familial Hypercholesterolemia or Familial Combined Hyperlipidemia
* Able to read, write and understand English
* Parental consent and child assent
* Access to a computer and internet and literacy in the use of the internet
* The attendance of a parent to each educational session.

Exclusion Criteria:

* Chronic systemic illness with or without secondary hyperlipidemia
* Current smoking

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2010-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Endothelial function | Measured every 6 wks for 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marguerite M. Engler, PhD, Principal Investigator — University of California, San Francisco; Mary B. Engler, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States